CLINICAL TRIAL: NCT02796794
Title: Effect of Enteral Genistein Supplementation on Inflammatory Cytokines, Morbidity and Mortality in Patients With Sepsis
Brief Title: Effect of Enteral Genistein Supplementation in Sepsis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Kursat Gundogan, MD, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/341
Record Dates: First submitted 2016-03-10; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Sepsis
Keywords: Enteral nutrition; Genistein; Cytokine
MeSH Terms: conditions — Sepsis | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genistein (Active Comparator): Intervention group will receive supplemental genistein (60 mg/day) to enteral nutrition
  Interventions: Dietary Supplement: Genistein
- control (Other): Control group are the patients receiving enteral nutrition
  Interventions: Other: enteral nutrition only

INTERVENTIONS:
Dietary Supplement: Genistein — Total 30 patients will be included into the study They will be divided into two groups each containing 15 patients. Intervention group will receive supplemental genistein (60 mg/day) to enteral nutrition
  Arms: Genistein
Other: enteral nutrition only — These are the patients receiving enteral nutrition
  Arms: control

SUMMARY:
To evaluate effects of genistein supplementation to enteral nutrition on inflammatory cytokines and morbidity in patients with sepsis

DETAILED DESCRIPTION:
Sepsis is a state develops as a response to severe infection with high mortality rate. Incidence of sepsis among patients admitted to hospitals is 2%. Annual incidence of sepsis is 50-95 for 100.000 population and incidence is increasing approximately 9% each year. Severe sepsis and septic shock is the most frequent reason for mortality in intensive care units (ICU). There is exaggerated and irregular host response in sepsis. Cytokines such as interleukin-1, interleukin-6, interleukin-8, tumor necrosis factor-α, Interferon-γ and high mobility group box-1 are released as response to invading microorganisms and they play a major role in sepsis pathogenesis.

Soybean proteins are used for prevention and treatment of cardiovascular diseases, osteoporosis and different cancer types.

Soy isoflavones such as genistein, daidzein and glycitein are the main components for cancer prevention. Genistein is the dominant isoflavones.

The main mechanism for anti-inflammatory effect of genistein is related to transcription nuclear factor (NF-kB) and inhibition of chemokine-8. The risk for prostate cancer was proven to decrease in epidemiological studies.

NF-kB plays a central role for inflammatory cytokine release, prevents apoptosis and induces tumor cell growth. The effect of topoisomerase II inhibitory chemotherapeutic agents is increased with NF-kB inhibition.

Hypothesis

1. Addition of genistein to enteral nutrition in patients with sepsis can play an important role to decrease inflammatory cytokines.
2. Morbidity can be decreased with lower levels of inflammatory cytokines in patients with sepsis.

ELIGIBILITY:
Criteria: inclusion criteria:

* Patients with sepsis above 18 years of age.
* Expected duration of ICU survival more than 48 hours.
* Patients receiving enteral nutrition (EN)
* Sepsis diagnosis within first 12 hours

Exclusion Criteria:

* Presence of thyroid dysfunction
* Presence of hyperlipidemia
* Patients with nill by mouth and not receiving enteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in Tumor necrosis factor alpha serum levels | Baseline, at 24th hour and at 72nd hour
  It will be measured at baseline, at 24th hour and at 72nd hour after inclusion into the study
Change in interleukin 1-beta serum levels | Baseline, at 24th hour and at 72nd hour
  It will be measured at baseline, at 24th hour and at 72nd hour after inclusion into the study
Change in interleukin 6 serum levels | Baseline, at 24th hour and at 72nd hour
  It will be measured at baseline, at 24th hour and at 72nd hour after inclusion into the study
Change in high-mobility group box 1 serum levels | Baseline, at 24th hour and at 72nd hour
  It will be measured at baseline, at 24th hour and at 72nd hour after inclusion into the study

SECONDARY OUTCOMES:
Number of study participants with development of new pneumonia, urinary tract infection and blood stream infections | From date of randomization until 12 weeks
  Patients will be followed until they are discharged from the hospital or death.
Length of intensive care unit and hospital stay (days) | From date of randomization until 12 weeks
  Patients will be followed until they are discharged from the hospital or death.
Duration of mechanical ventilation | From date of randomization until 12 weeks
  Patients will be followed until they are discharged from the hospital or death.
Intensive care unit mortality rate, hospital mortality rate | From date of randomization until 12 weeks
  Patients will be followed until they are discharged from the hospital or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Medical School, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Souza LR, Silva E, Calloway E, Kucuk O, Rossi M, McLemore ML. Genistein protects hematopoietic stem cells against G-CSF-induced DNA damage. Cancer Prev Res (Phila). 2014 May;7(5):534-44. doi: 10.1158/1940-6207.CAPR-13-0295. Epub 2014 Mar 10. PMID 24614013
- [Background] Lazarevic B, Hammarstrom C, Yang J, Ramberg H, Diep LM, Karlsen SJ, Kucuk O, Saatcioglu F, Tasken KA, Svindland A. The effects of short-term genistein intervention on prostate biomarker expression in patients with localised prostate cancer before radical prostatectomy. Br J Nutr. 2012 Dec 28;108(12):2138-47. doi: 10.1017/S0007114512000384. Epub 2012 Mar 8. PMID 22397815
- [Background] Hong H, Landauer MR, Foriska MA, Ledney GD. Antibacterial activity of the soy isoflavone genistein. J Basic Microbiol. 2006;46(4):329-35. doi: 10.1002/jobm.200510073. PMID 16847837
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731